CLINICAL TRIAL: NCT03373617
Title: The Effect of Anesthesia Type on the Surgical Field in Retrograde Intrarenal Surgery With Flexible Ureteroscopy in Renal Stone Patients
Brief Title: The Effect of Anesthesia Type on RIRS
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jung-Man Lee, Clinical assistant professor, Seoul National University Hospital
Other Study IDs: 20-2017-10
Record Dates: First submitted 2017-12-11; First posted 2017-12-14 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Renal Stone
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General anesthesia group: Patients in general anesthesia group are scheduled to undergo RIRS under general anesthesia.
- Spinal anesthesia group: Patients in spinal anesthesia group are scheduled to undergo RIRS under spinal anesthesia

SUMMARY:
Retrograde intrarenal surgery (RIRS) with flexible ureteroscopy is based on video monitoring of urinary tract during operation. Therefore, shaking vision on monitor can bother surgeons and make them tired. This can lead in tissue injury from lasing.

The purpose of this study is to investigate the stability of monitoring of surgical field which is assessed by surgeon.

DETAILED DESCRIPTION:
RIRS with flexible ureteroscopy is usually performed under general anesthesia, spinal anesthesia.

Anesthesia type is decided in the basis of medical condition of a patient and patient's preference.

This study is a prospective observational study. During operation after induction of anesthesia, surgeons will be asked how visual stability of surgical field on monitor is (scale from 0 to 10).

According to anesthesia type (general anesthesia, spinal anesthesia), 34 patients will be enrolled and investigated in each group.

Investigators will compare the scale for visual stability of surgical field during RIRS.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring RIRS because of renal stone.

Exclusion Criteria:

* disagreement for the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring RIRS because of renal stone
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2019-01-14 (Actual)

PRIMARY OUTCOMES:
VAS for stability of monitoring | intraoperative
  VAS (from 1 to 10) for stability in monitoring of surgical field, which is assessed by surgeons

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Man Lee, M.D.,PhD, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul, South Korea